CLINICAL TRIAL: NCT02636712
Title: Observation of ImageReady™ MR Conditional Pacing System in China
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C1913
Record Dates: First submitted 2015-12-11; First posted 2015-12-22 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-01

CONDITIONS: Arhythmia; Atrioventricular Heart-block; Chronic Bundle Branch or Branch Block; Carotid Sinus Hypersensitivity Reaction Syndrome; Vasovagal Syncope
MeSH Terms: conditions — Atrioventricular Block; Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ImageReady™ MR Conditional Pacing System: 1. Subject must have the ImageReady™ System as their initial (de novo) pacing system implant
  2. Subject has a Class I or II indication for implantation of a pacemaker according to the CSPE guidelines
  Interventions: Device: ImageReady™ MR Conditional Pacing System

INTERVENTIONS:
Device: ImageReady™ MR Conditional Pacing System

SUMMARY:
To observe the safety and efficacy of ImageReady™ MR Conditional Pacing System in Chinese subjects

DETAILED DESCRIPTION:
Key Inclusion Criteria:

1. Subject must have the Image Ready System as their initial (de novo) pacing system implant.
2. Subject has a Class I or II indication for implantation of a pacemaker according to the CSPE guidelines.
3. Subject is able and willing to undergo an MR scan.•
4. Subject is willing and capable of providing informed consent and participating in all testing/ visits associated with this clinical study at the intervals defined by this protocol.
5. Subject is age 18 or above.

Key Exclusion Criteria

1. Subject has or has had any pacing or ICD system implants.
2. Subject has any implants or devices that are not suitable for MR scan.
3. Subject is enrolled in any other concurrent study that might interfere with this study.
4. Subject has documented life expectancy of less than 12 months.
5. Women of childbearing potential who are or might be pregnant at the time of this study.

Primary Safety Endpoint:

MR Scan related Complication Free Rate Analyzed at MRI Visit +1 Month.

Primary efficacy Endpoint:

1. Pacing Threshold (at 0.5 ms pulse width) comparison pre and 1 Month post MR Scan: pacing threshold increase ≤ 0.5 V after scan.
2. Sensed Amplitude comparison pre- and 1 Month post-MR Scan: sensed amplitude: ≥ 1.0 mV after scan, and ≥ 50% of that before scan.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ImageReady System as their initial (de novo) pacing system implant
* Subject has a Class I or II indication for implantation of a pacemaker according to the CSPE guidelines5
* Subject is able and willing to undergo an MR scan
* Subject is willing and capable of providing informed consent and participating in all testing/ visits associated with this clinical study at the intervals defined by this protocol
* Subject is age 18 or above

Exclusion Criteria:

* Subject has or has had any pacing or ICD system implants
* Subject has any implants or devices that are not suitable for MR scan
* Subject is enrolled in any other concurrent study that might interfere with this study
* Subject has documented life expectancy of less than 12 months
* Women of childbearing potential who are or might be pregnant at the time of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in the MR China Study should be selected from the investigator's general patient population indicated for single or dual chamber pacemaker implantation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yangang Su, Doctor, Principal Investigator — Shanghai Zhongshan Hospital; Kejiang Cao, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nazarian S, Hansford R, Roguin A, Goldsher D, Zviman MM, Lardo AC, Caffo BS, Frick KD, Kraut MA, Kamel IR, Calkins H, Berger RD, Bluemke DA, Halperin HR. A prospective evaluation of a protocol for magnetic resonance imaging of patients with implanted cardiac devices. Ann Intern Med. 2011 Oct 4;155(7):415-24. doi: 10.7326/0003-4819-155-7-201110040-00004. PMID 21969340
- [Background] Russo RJ. Determining the risks of clinically indicated nonthoracic magnetic resonance imaging at 1.5 T for patients with pacemakers and implantable cardioverter-defibrillators: rationale and design of the MagnaSafe Registry. Am Heart J. 2013 Mar;165(3):266-72. doi: 10.1016/j.ahj.2012.12.004. Epub 2013 Jan 28. PMID 23453091
- [Background] BSC data on file. 91022242_SAMURAI_FDA endpoint report_29JUN2015_Final_revAC.
- [Background] ASTM Standard F2503-08, "Standard Practice for Marking Medical Devices and Other Items for Safety in the Magnetic Resonance Environment" ASTM International, West Conshohocken, PA, 2008, DOI: 10.1520/F2503-08, www.astm.org
- [Background] Wolf SM, Lawrenz FP, Nelson CA, Kahn JP, Cho MK, Clayton EW, Fletcher JG, Georgieff MK, Hammerschmidt D, Hudson K, Illes J, Kapur V, Keane MA, Koenig BA, Leroy BS, McFarland EG, Paradise J, Parker LS, Terry SF, Van Ness B, Wilfond BS. Managing incidental findings in human subjects research: analysis and recommendations. J Law Med Ethics. 2008 Summer;36(2):219-48, 211. doi: 10.1111/j.1748-720X.2008.00266.x. PMID 18547191
- [Background] Kanal E, Barkovich AJ, Bell C, Borgstede JP, Bradley WG Jr, Froelich JW, Gilk T, Gimbel JR, Gosbee J, Kuhni-Kaminski E, Lester JW Jr, Nyenhuis J, Parag Y, Schaefer DJ, Sebek-Scoumis EA, Weinreb J, Zaremba LA, Wilcox P, Lucey L, Sass N; ACR Blue Ribbon Panel on MR Safety. ACR guidance document for safe MR practices: 2007. AJR Am J Roentgenol. 2007 Jun;188(6):1447-74. doi: 10.2214/AJR.06.1616. No abstract available. PMID 17515363
- [Background] 张澍, 华伟, 黄德嘉, 王景峰, 吴立群, 杨杰孚, 曹克将, 黄从新, 王方正, 陈新: 植入性心脏起搏器治疗--目前认识和建议(2010年修订版). 中华心律失常学杂志 2010; 04:245-249. Shu Zhang, Wei Hua, Dejia Huang, Jingfeng Wang, Liqun Wu, Jiefu Wu, Kejiang Cao, Congxin Huang, Fangzheng Wang, Xin Chen: Implantable Cardiac Pacemaker therapy- Cognition and Suggestion Present ( updated version on 2010). Chinese Journal of Cardiac Arrhythmia, 2010; 04:245-249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment has finished on 25 Dec 2015 and totally 10 patients.
Groups:
- ImageReady™ System Indication: 1. Subject must have the ImageReady™ System as their initial (de novo) pacing system implant
  2. Subject has a Class I or II indication for implantation of a pacemaker according to the CSPE guidelines
  ImageReady™ MR Conditional Pacing System
Period: Overall Study
Arm/Group | ImageReady™ System Indication
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ImageReady™ System Indication
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: Year] | 69.4 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  China | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Complications at MRI Visit + 1 Month.
Description: No one has any complications related MR Scan . So Complication-Free rate is 100%.
Time Frame: Within 1 month after the Pacemaker been implanted.
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Groups:
- ImageReady™ MR System Indication: 1. Subject must have the ImageReady™ System as their initial (de novo) pacing system implant
  2. Subject has a Class I or II indication for implantation of a pacemaker according to the CSPE guidelines
  ImageReady™ MR Conditional Pacing System
Arm/Group | ImageReady™ MR System Indication
Number analyzed (Participants) | 10
percentage of paticipants | 100 [69.2 to 100]

2. Primary Outcome: Percentage of Participants Reporting an Increase in Pacing Thresholds ≤ 0.5V (at 0.5 ms) From Pre-MR Scan to MRI Visit + 1 Month Follow-up
Description: The percentage of Participants Reporting an Increase in Pacing Thresholds ≤ 0.5V (at 0.5 ms) from Pre-MR Scan to MRI Visit + 1 Month Follow-up is 100 percent.
Time Frame: Pre-MR scan and 1 Month post-MR Scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ImageReady™ System Indication
Number analyzed (Participants) | 10
percentage of participants | 100 [80.5 to 100]

3. Primary Outcome: Percentage of Participants With Atrial Sensed Amplitude at the MRI Visit + 1 Month Follow up Remains ≥ 1.0 mV and Above 50% of the Pre-MR Scan Value
Description: The Percentage of participants with atrial sensed amplitude at the MRI Visit + 1 Month Follow up remains ≥ 1.0 mV and above 50% of the pre-MR scan value is 100%.
Time Frame: Pre-MR scan and 1 Month post-MR Scan.
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | ImageReady™ System Indication
Number analyzed (Participants) | 10
percentage of paticipants | 100 [59 to 100]

4. Primary Outcome: Percentage of Participants With Ventricular Sensed Amplitudes at the MRI Visit + 1 Month Follow up Remains ≥ 5.0 mV and Above 50% of the Pre-MR Scan.
Description: The percentage of participants with ventricular sensed amplitudes at the MRI Visit + 1 Month Follow up remains ≥ 5.0 mV and above 50% of the pre-MR scan is 100%.
Time Frame: Pre-MR scan and 1 Month post-MR Scan.
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | ImageReady™ System Indication
Number analyzed (Participants) | 10
percentage of paticipants | 100 [69.2 to 100]

5. Secondary Outcome: Percentage of Participants Without System-related Complications
Description: No one has any complications related system occurred. So Complication-Free rate is 100%.
Time Frame: Within 3 months after the Pacemaker been implanted.
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | ImageReady™ System Indication
Number analyzed (Participants) | 10
percentage of paticipants | 100 [69.2 to 100]

ADVERSE EVENTS:
Time Frame: Pre-Discharge, MR Scan Visit, MRI Visit+1 Week, MRI Visit+1 Month
Groups:
- ImageReady™ MR Conditional Pacing System: 1. Subject must have the ImageReady™ System as their initial (de novo) pacing system implant
  2. Subject has a Class I or II indication for implantation of a pacemaker according to the CSPE guidelines
  ImageReady™ MR Conditional Pacing System
Arm/Group | ImageReady™ MR Conditional Pacing System
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady™ MR Conditional Pacing System (N=10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ImageReady™ MR Conditional Pacing System (N=10)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes